CLINICAL TRIAL: NCT00692887
Title: Correlation Between Visual Field Defects on Foresee PHP and OCT in Patients With CNV Before and After Treatment
Brief Title: Correlation Between Visual Field Defects on Foresee Preferential Hyperacuity Perimeter(PHP) and on Optical Coherence Tomography (OCT) in Patients With Choroidal Neovascularization (CNV)
Acronym: PHP
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Osnat Ehrman, Notal Vision
Organization: Notal Vision Inc. (Industry)
Other Study IDs: PHP-POST-01
Record Dates: First submitted 2008-05-26; First posted 2008-06-06 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Subjects diagnosed as new CNV or treated CNV
  Interventions: Device: PHP - Preferential Hyperacuity Perimeter (Foresee)

INTERVENTIONS:
Device: PHP - Preferential Hyperacuity Perimeter (Foresee) — computerized test
  Other Names: PHP 2.0.5; OCT - optical coherence tomography

SUMMARY:
Study come to investigate the correlation between visual fields (VF) defects map generated by preferential hyperacuity perimeter (PHP) and features of the choroidal neovascular lesions (CNV) demonstrated by Optical Coherence Tomography(OCT).

To investigate the Foresee PHP ability to asses treatment progression post treatment.

DETAILED DESCRIPTION:
The Foresee PHP is used in the recent years to detect Age-related Macular Degeneration (AMD) lesions. The device is capable of differentiation as to stages of AMD and early detection of changes including choroidal neovascularization (CNV) The Foresee PHP™ demonstrates a high level of sensitivity and specificity as to the different stages of AMD including newly diagnosed or early detection of CNV.

The OCT May be use as well to identify choroidal neovascularization (CNV). Comparison between the two methods will allow better understanding of both devices.

The Foresee PHP can use as an assessment tool for the progression and success of the treatment given to AMD lesions. Therefore, evaluation the size and the location of the treated lesions may serve as an additional tool.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study
* Subjects diagnosed as new CNV or treated CNV
* Age >50 years
* VA with habitual correction <20/160 in the study eye
* Ability to understand instructions

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy,
* Any non-macular related ocular surgery performed within 3 months prior to study entry in the target eye
* Patients diagnosed with geographic atrophy (GA)
* Participation in another study with the exclusion of AREDS study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Subjects diagnosed as new CNV or treated CNV
  * Age >50 years
  * VA with habitual correction <20/160 in the study eye
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To investigate the correlation between visual fields (VF) defects map generated by preferential hyperacuity perimeter (PHP) and features of the choroidal neovascular lesions (CNV) demonstrated by Optical Coherence Tomography(OCT). | 6 month

SECONDARY OUTCOMES:
To investigate the Foresee PHP ability to asses treatment progression post treatment. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Anat Loewenstein, Prof., Principal Investigator — Sorasky Medical Center
Locations (1):
- Sorasky Medical center, Tel Aviv, Israel

REFERENCES:
- See also: sponsor web site — http://www.notalvision.com